CLINICAL TRIAL: NCT06253767
Title: Analysis of Post-Endodontic Instrumentation Pain in Molars and Premolars Treated in a Single Session Associated With Photobiomodulation: A Double-blind Randomized Clinical Study
Brief Title: Post-Endodontic Instrumentation Pain After in a Single Session Associated With Photobiomodulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Principal investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5991.5622.3.0000.5511
Record Dates: First submitted 2024-01-05; First posted 2024-02-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pain, Postoperative; Endodontically Treated Teeth
Keywords: photobiomodulation; analgesia
MeSH Terms: conditions — Pain, Postoperative; Tooth, Nonvital; Agnosia | interventions — Endodontics; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (TG) (Experimental): They are composed of 29 participants. After endodontic treatment, they will receive PBM for molars with 808nm application (AsGaAl), infrared, equipment with a power of 100 mW, and an exit beam area of 1 cm² perpendicular in contact with the mucosa at the level of the root apices at two vestibular points and one complementary palatal point, with 3J of energy per point (30s per point), totaling 9J of total delivered energy and 90 seconds of application time. The Radiant Exposure is 3J/cm² per point, totaling 9J/cm² overall. To premolars the parameters will be 808nm application (AsGaAl), infrared, Laser Duo® equipment with a power of 100 mW and an exit beam area of 1cm² perpendicular in contact with the mucosa at the level of the root apices at one vestibular point and one complementary palatal point, with 3J of energy per point (30s per point), totaling 6J of total delivered energy and 60 seconds of application time. The Radiant Exposure is 3J/cm² per point, totaling 6J/cm² overall
  Interventions: Procedure: Endodontic Treatment; Device: Low Level Laser Therapy
- Control Group (CG) (Sham Comparator): They are composed of 29 participants. After endodontic treatment, they will receive a simulation of the PBM session with all individual preparation involved, such as individual protection with goggles, and the sounds of the equipment (Laser Duo®, MMOptics, São Carlos, SP) will be recorded and played at the time of the session, but the equipment will not be activated.
  Interventions: Procedure: Endodontic Treatment; Device: Simulation Low Level Laser therapy

INTERVENTIONS:
Procedure: Endodontic Treatment — Conventional endodontic treatment will be performed equally on all participants.
Device: Low Level Laser Therapy — Treatment Group (TG) will receive photobiomodulation for molars with 808nm application (AsGaAl), infrared, equipment with a power of 100 mW, and an exit beam area of 1 cm² perpendicular in contact with the mucosa at the level of the root apices at two vestibular points and one complementary palatal point, with 3J of energy per point (30s per point), totaling 9J of total delivered energy and 90 seconds of application time. The Radiant Exposure is 3J/cm² per point, totaling 9J/cm² overall. To premolars the parameters will be 808nm application (AsGaAl), infrared, Laser Duo® equipment with a power of 100 mW and an exit beam area of 1cm² perpendicular in contact with the mucosa at the level of the root apices at one vestibular point and one complementary palatal point, with 3J of energy per point (30s per point), totaling 6J of total delivered energy and 60 seconds of application time. The Radiant Exposure is 3J/cm² per point, totaling 6J/cm² overall
  Arms: Treatment Group (TG)
Device: Simulation Low Level Laser therapy — A simulation of low-level laser therapy was performed on the control group starting from patient preparation (placement of glasses) and the reproduction of device sounds without activation.
  Arms: Control Group (CG)

SUMMARY:
The objective of this double-blind, randomized controlled clinical study will be to evaluate the effect f PBM on pain after endodontic instrumentation in the single-session treatment of upper molars and premolars. The sample will consist of 58 participants treated endodontically in a single session and randomly allocated to the PBM Group with conventional treatment with photobiomodulation and the Control Group with conventional treatment with simulation of PBM. The primary variable of the study will be the evaluation of spontaneous pain immediately before treatment, and the participant will be reassessed for postoperative pain 24 hours after instrumentation using the visual analog scale (VAS). As secondary variables, pain prevalence, pain at 4h, 8h, and 12h after the procedure, palpation pain (vestibular and lingual), and percussion pain (vertical and horizontal) will be assessed 24 hours after the procedure, as well as the number of necessary analgesics (paracetamol) and the impact of oral health on quality of life evaluated by the OHIP 14 instrument.

DETAILED DESCRIPTION:
The randomized clinical trials conducted in recent years have demonstrated that photobiomodulation (PBM) modulates postoperative pain in endodontic instrumentation, especially in the first days after the procedure. Although the results are promising, there is still low-quality evidence regarding the best dosimetric parameter applied. The objective of this double-blind, randomized controlled clinical study will be to evaluate the effect of PBM on pain after endodontic instrumentation in the single-session treatment of upper molars and premolars. The sample will consist of 58 participants treated endodontically in a single session and randomly allocated to the PBM Group (n=29): conventional treatment with photobiomodulation (808 nm, 100mW power, 3J per point, 3mm2 area, 3 points in the region of the root apices - two vestibular and one palatal, total energy of 9J - for molars and premolars 2 points - 1 vestibular and another palatal, total energy of 6J) and Control Group (n=29): conventional treatment with simulation of PBM. The primary variable of the study will be the evaluation of spontaneous pain immediately before treatment, and the participant will be reassessed for postoperative pain 24 hours after instrumentation using the visual analog scale (VAS). As secondary variables, pain prevalence, pain at 4h, 8h, and 12h after the procedure, palpation pain (vestibular and lingual), and percussion pain (vertical and horizontal) will be assessed 24 hours after the procedure, as well as the number of necessary analgesics (paracetamol) and the impact of oral health on quality of life evaluated by the OHIP 14 instrument.

ELIGIBILITY:
Inclusion Criteria:

* Patients with endodontic involvement in three-rooted (upper molars) or two-rooted (upper premolars) teeth.
* Age between 20 and 75 years.
* Both genders.

Exclusion Criteria:

* Pregnancy or lactation.
* Patients with oncological, renal, or Type I or Type II diabetes.
* Drug users; alcohol or tobacco users.
* Immunocompromised patients or those using immunosuppressive medication.
* Use of alendronate, bisphosphonates, or any systemic medication that interferes with bone metabolism.
* Presence of associated periodontal disease.
* Frequent exacerbations.
* Radiolucency images with PAI stages 3, 4, or 5 (Orstavik et al., 1986).
* Any other anatomical variation that renders single-session endodontic treatment unfeasible.
* Teeth with previous endodontic treatment.
* Patients with asymptomatic non-microbial apical periodontitis with any type of bruxism (clenching) or using a bite splint.
* Teeth with more than ⅔ coronal involvement, making proper use of rubber dam isolation impossible.
* Use of antibiotics in the last three months.
* History of severe allergy to chlorine or its derivatives.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Baseline : Analysis of pain before treatment | Immediately before the treatment
  Before the treatment, regardless of the patient's randomized group, pain assessment will be conducted on the tooth and the surrounding area through palpation and percussion exams. Therefore, the patient will mark on the visual pain scale corresponding to their immediate pain, pain upon palpation, and pain upon percussion just before the treatment. The researcher will measure, using a ruler, the distance from "0" (no pain) to the patient's marked point, and this value will be taken as the comparator.
Analysis of Postoperative Pain at 4 Hours After Treatment | 4 hours after treatment
  After root canal obturation, all participants will receive a sheet containing a visual pain scale to document postoperative pain at 4 hours after the procedure. This scale will be exactly 10 cm and will range from 0 to 10, where the participant must mark a level representing their pain at that moment. This mark will be measured with a ruler, and the corresponding level will be noted.
Analysis of Postoperative Pain at 8 Hours After Treatment | 8 hours after treatment
  After root canal obturation, all participants will receive a sheet containing a visual pain scale to document postoperative pain at 8 hours after the procedure. This scale will be exactly 10 centimeters and will range from 0 to 10, where the participant must mark a level representing their pain at that moment. This mark will be measured with a ruler, and the corresponding level will be noted.
Analysis of Postoperative Pain at 12 Hours After Treatment | 12 hours after treatment
  After root canal obturation, all participants will receive a sheet containing a visual pain scale to document postoperative pain at 12 hours after the procedure. This scale will be exactly 10 centimeters and will range from 0 to 10, where the participant must mark a level representing their pain at that moment. This mark will be measured with a ruler, and the corresponding level will be noted.
Analysis of Postoperative Pain at 24 Hours After Treatment | 24 hours after treatment
  24 hours after the root canal filling, whether or not accompanied by photobiomodulation, the patient will return to the clinic for a reassessment of immediate pain. At this moment, the patient will be provided with a visual analog scale consisting of exactly 10 centimeters, with markings of "0" (no pain) and "10" representing maximum pain. The patient will then make a mark on this scale to indicate their current level of pain in the dental element. After the marking, the researcher will measure the distance from zero to the marked point using a millimeter ruler, and the obtained result will be recorded and statistically compared with the preoperative pain.

SECONDARY OUTCOMES:
Baseline : Analysis of pain upon palpation before treatment | Immediately before the treatment
  Before the treatment, regardless of the patient's randomized group, pain assessment will be conducted on the tooth and the surrounding area through palpation and percussion exams. Therefore, the patient will mark on the visual pain scale corresponding to their immediate pain, pain upon palpation, and pain upon percussion just before the treatment. The researcher will measure, using a ruler, the distance from "0" (no pain) to the patient's marked point, and this value will be taken as the comparator.
Analysis of Palpation Pain 24 Hours After Treatment | 24 hours after treatment
  During the same follow-up appointment 24 hours after endodontic treatment, palpation pain (vestibular and palatal) will be analyzed. The participant, after palpating the vestibular board, will mark on the visual pain scale the level of referred pain, and the same procedure will be done after palpating the palatal bony board.
Baseline: Analysis of pain upon percussion before treatment | Immediately before the treatment
  Before the treatment, regardless of the patient's randomized group, pain assessment will be conducted on the tooth and the surrounding area through palpation and percussion exams. Therefore, the patient will mark on the visual pain scale corresponding to their immediate pain, pain upon palpation, and pain upon percussion just before the treatment. The researcher will measure, using a ruler, the distance from "0" (no pain) to the patient's marked point, and this value will be taken as the comparator.
Analysis of Percussion Pain 24 Hours After Treatment | 24 hours after treatment
  Percussion pain (vertical and horizontal) will also be assessed 24 hours after treatment. These assessments will be performed by the principal investigator, who is blinded to the treatment administered and properly calibrated.
Analysis of the Required Analgesic Quantity | 24 hours after treatment
  Following the completion of endodontic treatment, all participants will be provided with 750mg Paracetamol tablets, and they will be instructed to take them in case of extreme pain. The quantity of analgesic intake should be noted on the sheet provided for recording pain experiences and returned during the 24-hour follow-up appointment.
Oral Health Impact Profile-14 | 24 hours after treatment
  The effects of treatment on participants' quality of life will be assessed using the patient-centered outcome measures from the Oral Health Impact Profile-14 (OHIP-14). The questionnaire will be handed to participants at the end of the treatment, and they will be properly instructed to fill it out and return it during the 24-hour follow-up.
Prevalence Analysis | 24 hours after treatment
  In the prevalence analysis of a particular condition, the frequency of occurrence of the condition, or in this case, the painful condition, in a specific population at a single point in time or a short period will be obtained (Bonita et al., 1993). In this study, the prevalence of pain before and 24 hours after endodontic instrumentation in the single-session treatment of upper molars will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Carolina RT Horliana, Study Chair — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil